CLINICAL TRIAL: NCT04516226
Title: Vaginal Cleansing With Chlorhexidine Gluconate in Women With Preterm Pre-labor Rupture of Membranes in Order to Prolong Pregnancy Latency and Reduce Intraamniotic Inflammation
Brief Title: Vaginal Cleansing With Chlorhexidine Gluconate in Women With Preterm Pre-labor Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5743
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal cleansing (Experimental): This group includes patients diagnosed with PPROM that are randomized to undergo vaginal cleansing with chlorhexidine gluconate within 24 hours of PPROM diagnosis.
  Interventions: Other: Vaginal cleansing with chlorhexidine gluconate solution
- No vaginal cleansing (No Intervention): This group includes patients diagnosed with PPROM that are randomized to not undergo vaginal cleansing.

INTERVENTIONS:
Other: Vaginal cleansing with chlorhexidine gluconate solution — Cleansing of the vaginal walls with chlorhexidine gluconate solution for women diagnosed with PPROM
  Arms: Vaginal cleansing

SUMMARY:
Randomized controlled trial studying the use of vaginal cleansing with chlorhexidine gluconate for pregnant women with PPROM (preterm pre labor rupture of membranes). The primary outcome will be pregnancy latency. Secondary outcomes will include various maternal and neonatal outcomes, and inflammatory markers from maternal blood, amniotic fluid, fetal cord blood and placental analysis.

DETAILED DESCRIPTION:
A randomized controlled trial, including pregnant women > 18 years old with early onset PPROM occurring between the time of peri-viability through the early third trimester (20 weeks 0 days - 33 weeks 0 days) at Albany Medical Center.

Women will be consented by a physician member of the research team on labor and delivery after clinical diagnosis of PPROM. Participation will be completely voluntary and not impact routine prenatal care for PPROM, which may include but not be limited to hospital admission, standard latency antibiotics, NICU consultation, fetal growth ultrasounds, fetal monitoring, and delivery will be based on physician assessment and not impacted by this study. Participation in the study will involve prospective data collection on maternal, fetal, and neonatal characteristics, randomization into a control and treatment group, collection of maternal serum, fetal cord blood and vaginal fluid. Subjects will be randomized into control and treatment groups via block randomization. Exclusions will include any contraindications to expectant management for PPROM noted at the time on admission, such as preterm labor, chorioamnionitis, maternal sepsis and fetal distress.

The time commitment for each subject will include the time from diagnosis of PPROM until their delivery. Although outcome measures will be collected from each neonate, no further participation from subjects will be required after time of their delivery.

Treatment Group: Women diagnosed with PPROM (20 - 33 weeks) randomized to the treatment group will undergo vaginal cleansing with chlorhexidine gluconate within 24 hours of their diagnosis. This specific procedure will only be done once.

The vaginal cleansing procedure will be performed by a single investigator, Dr. Cagino, to ensure consistency. The patient will be examined in dorsal lithotomy position with a standard speculum. A sterile 2x2 gauze placed on ringed forceps will be soaked in sterile 2% chlorhexidine gluconate in

aqueous solution (all available on labor and delivery). Only the rough volume of 2% chlorhexidine gluconate required to soak the small sterile gauze will be used. This soaked gauze will be used to carefully wipe the vaginal mucosa of the vaginal vault. No pooling of chlorhexidine will be left in the vaginal vault. The chlorhexidine solution will not be applied to the cervix or cervical os. The chlorhexidine solution will not be applied directly to the fetus in any way. If a fetal part is visualized at time of exam, the patient will be excluded from the study.

Otherwise, standard care for PPROM among women in this group will not change. This group will be expectantly managed until the time of delivery, which will be based on physician assessment. Delivery decisions for women with preterm labor or infection will be based on physician assessment only and will not be influenced by their involvement in this study.

Control Group: Women diagnosed with PPROM (20 - 33 weeks) randomized to the control group will undergo standard care for PPROM. This group will be expectantly managed until the time of delivery, which will be based on physician assessment. Data will be collected from both the patient and neonate (please see the collection sheet for further information).

Inclusions:

* Pregnant patients at Albany Medical Center with PPROM diagnosed between 20 - 33 weeks
* Age > 18 years old

Exclusions:

* Active preterm labor or imminent delivery expected at time of PPROM diagnosis
* Maternal sepsis or chorioamnionitis diagnosed at time of PPROM diagnosis
* Any contraindications to expectant management at time of PPROM diagnosis (fetal distress, placental abruption with maternal hemodynamic instability or fetal distress, cord prolapse)
* Preeclampsia
* Intrauterine growth restriction (IUGR)
* No antibiotics or steroids given within 7 days prior to time of enrollment/randomization in study (not including steroids or treatment given during admission)
* Multiple gestation
* Placenta previa
* Fetal part visualized at initial exam
* Visual cervical dilation at initial exam

Primary Outcome: Latency (days from PPROM to delivery)

Secondary Outcomes:

* Serum IL6, IL10, TNF-a - admission, day 7, delivery
* Vaginal fluid IL6, IL10, TNF-a - admission, day 7, delivery
* Serial antepartum CBC - admission, day 7, delivery
* Postpartum CBC
* Clinical chorioamnionitis (as defined by treating clinician discretion and requiring treatment with antibiotics and/or delivery)
* Placenta pathology (per pathology lab)
* Histologic chorioamnionitis (based on placental pathology)
* Maternal sepsis (as defined by treating clinician discretion)

  * Culture proven
  * Presumed sepsis
* Composite neonatal morbidity
* Neonatal death
* Fetal demise

A power analysis was performed based on the mean latency of 18 days (SD 10 days) in patients who remained pregnant at least 7 days following PPROM at AMC. In order to detect a prolongation in latency by at least 10 days in the treatment group, an effect size of 1, with a power 0.8 and alpha 0.05, 17 subjects in each study group are needed. A study duration of 1.5 to 2 years to complete enrollment, data collection and analysis is anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients at our institution with PPROM diagnosed between 20 - 33 weeks

Exclusion Criteria:

* active preterm labor or imminent delivery expected at the time of PPROM diagnosis
* maternal sepsis or chorioamnionitis
* any contraindications to expectant management (fetal distress, placental abruption with maternal hemodynamic instability or fetal distress cord prolapse)
* preeclampsia
* intrauterine growth restriction (IUGR)
* no antibiotics or steroids given within 7 days prior to the time of enrollment
* multiple gestation
* placenta previa
* fetal part visualized at initial exam
* visual cervical dilation at initial exam

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy latency | Delivery
  The time measured in days from the diagnosis of pre labor premature rupture of membranes (PPROM) to delivery.

SECONDARY OUTCOMES:
Serum inflammatory markers | Within 24 hours of admission, 7 days after admission, day of delivery
  Inflammatory markers from maternal serum including IL6, TNF-a, IL10
Amniotic fluid inflammatory markers | Within 24 hours of admission, 7 days after admission, day of delivery
  Inflammatory markers from amniotic fluid including IL6, TNF-a, IL10
White blood cell count, cells per liter | Within 24 hours of admission, 7 days after admission, day of delivery
  Maternal CBC measured serially antepartum and postpartum
Number of participants with clinical chorioamnionitis | Through study completion, an average of 1 year
  as defined by treating clinical, requiring treatment with antibiotics and/or delivery
Rate of placental abnormalities on pathology evaluation | studied postpartum, up to 1 week
  Histopathology per pathology lab
Rate of histologic chorioamnionitis | studied postpartum, up to 1 week
  based on placental pathology
Rate of maternal sepsis | through study completion, up to 1 year
  as defined by treating clinical, culture proven or presumed
rate of composite neonatal morbidity | through study completion, up to 1 year
  culture proven sepsis, respiratory distress, necrotizing enterocolitis, intracranial hemorrhage
rate of neonatal death | through study completion, up to 1 year
  demise of neonate
fetal demise | through study completion, up to 1 year
  demise of fetus in-utero

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No